CLINICAL TRIAL: NCT03629093
Title: General Anesthesia Exposed Infants Neurodevelopment Investigation: a Multi-center Prospective Cohort Study United in Shanghai
Brief Title: Neurodevelopment of Infants Exposed to General Anesthesia: a Multi-center Investigation
Acronym: GENIUS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Huashan Hospital (Other)
Collaborators: Shanghai Children's Medical Center (Other); Children's Hospital of Fudan University (Other); Shanghai Children's Hospital (Other); Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other); Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Xiao-Yu Yang, MD, Doctor, Huashan Hospital
Other Study IDs: GENIUS
Record Dates: First submitted 2018-08-08; First posted 2018-08-14 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: General Anesthetics Toxicity; Neurodevelopment; Infant
Keywords: General anesthesia; Infant; Neurodevelopment; Postoperative; the Gesell Developmental Inventory
MeSH Terms: interventions — Anesthetics, General; Anesthesia, General

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Long-time anesthesia exposure: Infants receive general anesthetics longer than 3 hours in total.
  Interventions: Drug: General Anesthetics
- Short-time anesthesia exposure: Infants receive general anesthetics shorter than 3 hours in total.
  Interventions: Drug: General Anesthetics

INTERVENTIONS:
Drug: General Anesthetics — General anesthesia required for surgery procedures or diagnostic interventions using either intravenous or inhalation anesthetics, or both.
  Other Names: General anesthesia

SUMMARY:
Numerous preclinical evidence has confirmed that most commonly-used general anesthetics can affect neurodevelopment of young animals adversely, causing both structural defect of brain and cognitive impairment. However, it is unclear at present whether such effect would also occur to children exposed to general anesthesia in their early life. Several observational clinical studies and one interventional clinical trial indicated that short-time general anesthesia less than 80 minutes might be safe to cognitive development. Concerning long-time and/or multiple anesthesia exposure, some studies supported its association with long-term cognitive defects, while other studies did not. These studies are mainly retrospective or ambirectional researches. We have designed a prospective, multicenter cohort study to examine the neurodevelopment of infants exposed to anesthesia before age 2 in the first year after surgery, and compare the neurodevelopment status of infants exposed to anesthesia less than 3 hours and those more than 3 hours. The Gesell Developmental Inventory (GDI) and several neuropsychological testing batteries will be used. The anticipated outcome of the study will add reliable evidence from Asians to elucidate the relationship of anesthesia and long-term neurodevelopment of infants.

ELIGIBILITY:
Inclusion Criteria:

* Apgar score ≥ 8 at birth
* ASA level Ⅰ~Ⅲ
* Obtained written consent form from the infants' parents or guardians

Exclusion Criteria:

* Postmenstrual age ≤ 44 weeks, or postmenstrual age ≥ 144 weeks
* Severe cardiac, pulmonary, or neurologic disease
* Severe obstructive sleep apnea hypopnea syndrome
* History of dystocia and/or hypoxic ischemic encephalopathy
* Gestational age at birth ≤32 weeks
* Any known or suspected chromosomal abnormalities, abnormal development of vision or hearing, neurodevelopment retardation, or other known acquired or congenital abnormalities that might affect neurodevelopment
* Significant cardiovascular surgery, significant ENT surgery, or neurosurgery
* Malignant diseases that may reduce survival
* Taking part in other clinical trials in the last 3 months or at present

Ages: 4 Weeks to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Eligible infants scheduled for elective surgeries under general anesthesia will be recruited in six medical centers in Shanghai, China. The medical centers include Huashan Hospital Fudan University, Shanghai Children's Medical Center, Children's Hospital of Fudan University, Children's Hospital of Shanghai, Shanghai Tenth People's Hospital, and Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Change of the developmental quotient of the Gesell Developmental Inventory | From baseline before anesthesia to 1 year after anesthesia
  The Gesell Developmental Inventory has been translated into Chinese and standardized by the Beijing Children's Health Care Institute and the performance results are expressed as a developmental quotient (DQ).

SECONDARY OUTCOMES:
Change of the standardized score of the five domains of the Gesell Developmental Inventory | From baseline before anesthesia to 1 year after anesthesia
  The five behavioral domains are gross motor, fine motor, language, adaptive, and personal-social behaviors.
Change of the standardized score of the Social Maturity Scale | From baseline before anesthesia to 1 year after anesthesia
  The Social Maturity Scale includes six domains and 132 questions designed to be completed by the parents.

CONTACTS AND LOCATIONS:
Overall Officials: Ying-Wei Wang, M.D., Ph.D., Study Director — Huashan Hospital
Locations (1):
- Huashan Hospital Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Davidson AJ, Disma N, de Graaff JC, Withington DE, Dorris L, Bell G, Stargatt R, Bellinger DC, Schuster T, Arnup SJ, Hardy P, Hunt RW, Takagi MJ, Giribaldi G, Hartmann PL, Salvo I, Morton NS, von Ungern Sternberg BS, Locatelli BG, Wilton N, Lynn A, Thomas JJ, Polaner D, Bagshaw O, Szmuk P, Absalom AR, Frawley G, Berde C, Ormond GD, Marmor J, McCann ME; GAS consortium. Neurodevelopmental outcome at 2 years of age after general anaesthesia and awake-regional anaesthesia in infancy (GAS): an international multicentre, randomised controlled trial. Lancet. 2016 Jan 16;387(10015):239-50. doi: 10.1016/S0140-6736(15)00608-X. Epub 2015 Nov 4. PMID 26507180
- [Background] Graham MR. Clinical update regarding general anesthesia-associated neurotoxicity in infants and children. Curr Opin Anaesthesiol. 2017 Dec;30(6):682-687. doi: 10.1097/ACO.0000000000000520. PMID 28915132
- [Background] Sun LS, Li G, Miller TL, Salorio C, Byrne MW, Bellinger DC, Ing C, Park R, Radcliffe J, Hays SR, DiMaggio CJ, Cooper TJ, Rauh V, Maxwell LG, Youn A, McGowan FX. Association Between a Single General Anesthesia Exposure Before Age 36 Months and Neurocognitive Outcomes in Later Childhood. JAMA. 2016 Jun 7;315(21):2312-20. doi: 10.1001/jama.2016.6967. PMID 27272582
- [Background] Warner DO, Zaccariello MJ, Katusic SK, Schroeder DR, Hanson AC, Schulte PJ, Buenvenida SL, Gleich SJ, Wilder RT, Sprung J, Hu D, Voigt RG, Paule MG, Chelonis JJ, Flick RP. Neuropsychological and Behavioral Outcomes after Exposure of Young Children to Procedures Requiring General Anesthesia: The Mayo Anesthesia Safety in Kids (MASK) Study. Anesthesiology. 2018 Jul;129(1):89-105. doi: 10.1097/ALN.0000000000002232. PMID 29672337